CLINICAL TRIAL: NCT02814734
Title: Abdominal Compartment Syndrome : Diagnostic and Prognostic Value of CT Findings - a Prospective Study
Acronym: SCANAPIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/298
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Intra-Abdominal Hypertension; Abdominal Compartment Syndrome
Keywords: Intra-Abdominal Hypertension; Abdominal Compartment Syndrome; Round Belly Sign; Radiology; CT findings; Intensive Care
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Abdominal Compartment Syndrome (ACS) is a well known condition occuring in critically ill patients in intensive care units.

This syndrome features a sustained intra abdominal hypertension (IAH) above 20 mmHg and a multiple organ failure due to the raise of the intra abdominal pressure.

Several reviews described CT findings linked to these conditions, but most of them suffer an insufficient statistical method.

Furthermore, the main CT feature described as specific in ACS, Round Belly Sign (RBS), has been highly debated since.

This study is aimed to evaluate, in a prospective way, the diagnostic and prognostic value of CT findings in abdominal hypertension and abdominal compartment syndrome patients hosted in intensive care units, based on previous reviews and adding three new CT features described for the first time.

DETAILED DESCRIPTION:
Abdominal compartment syndrome (ACS) is a well known condition, occurring in patients hosted in intensive care units and suffering from acute abdominal disease (such as severe acute pancreatitis, trauma, hemoperitoneum, surgery, infectious disease), large volume fluid resuscitation (over 2,5L), and systemic disease such as severe sepsis or major burns.

This syndrome features a sustained intra abdominal hypertension (IAH) above 20 mmHg, measured indirectly by intra-vesical pressure, and a multiple organ failure due to the raise of the intra abdominal pressure.

IAH, which is defined as an abdominal pressure rise above 12 mmHg, does not systematically lead to ACS, and is often successfully cured with medical therapy.

When medial management fails, or ACS is present, surgical management is appropriate and consists in a decompressive laparotomy.

CT examination is not ordered for ACS diagnostic, but radiologists should be aware of this condition and CT findings in patients with IAH, as these critically ill patients are likely to have multiple CT examinations in a diagnostic purpose for the initial condition, its complications or its surveillance.

Several radiological studies have determined CT findings of IAH and ACS. Most of them failed to establish a specific and sensitive semiology of IAH, due to weak methodology (except Al-Bahrani and al.). The diagnostic significance of the "Round Belly Sign" (RBS), first described by Pickhardt and al., has been debated since. None of these studies evaluated the prognostic value of IAH CT findings.

Some of IAH CT findings may have a prognostic value, and being statistically linked to a raised risk of ACS overcome when found in at-risk patients population, with proven IAH.

The aim of this study is to evaluate diagnostic and prognostic value of CT findings in IAH in a prospective way, with a high statistic value.

These CT findings are the ones previously described in previous reviews (round belly sign, narrowing of abdominal veins, elevation of the diaphragm, bilateral inguinal herniation, bowel wall thickening with enhancement, direct visceral compression) and the ones studied here for the first time (increase of the peritoneal/abdominal ratio, semi-lunar line distension, concavity of the upper side of the para renal fascia).

Design:

For each included patient, when an abdominal CT is ordered, an intra-abdominal pressure measure is performed simultaneously to the CT examination. Presence or absence of IAH or ACS is noted.

Two radiologists (one junior and one senior specialized in abdominal emergencies imaging) review the CT examinations and note the presence or absence of the ten CT features studied, without knowing the intra-abdominal pressure value.

Patient follow-up:

* 5 days follow-up
* intra-abdominal pressure measurements
* Incidence of ACS from the time of inclusion to 28 days after.
* Evolution of organ failures
* Vital status at 28 days
* Medical and surgical therapy applied

Analysis:

* Diagnostic value of CT findings in IAH
* Prognostic value of CT findings in IAH, defining CT features statistically linked to ACS overcome, and mortality at 28 days

Prevalence of IAH is expected to be about 40 to 50% in patients in state of shock hosted in ICU. Among them, about 20% are expected to suffer from ACS.

Sensitivity of RBS in IAH is about 80% according to Al-Bahrani and al.. To evaluate the diagnostic value of RBS with (CI = [0,68 - 0,88]), 68 cases of IAH and about 140 patients included are needed.

Based on imaging habits in our center, length of this study is expected to be about 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring ICU hosting
* State of shock requiring vasopressive drugs
* State of shock requiring mechanical ventilation
* Abdominal CT examination ordered
* Intra abdominal pressure measurement

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Contraindication to urethral catheter
* Decompressive laparotomy before CT examination
* Absolute contraindication to CT enhancement agent
* Cystectomy
* Trusteeship/guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients hosted in intensive care units (ICU) in state of shock requiring vasopressive drugs, mechanical ventilation, in which an abdominal CT is ordered and performed with simultaneous intra abdominal pressure measurement.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Intra abdominal hypertension (HIA) | Within four hours before or after the abdominal CT examination
  Incidence of intra-abdominal hypertension in patients included, defined by the raise above 12 mmHg of the intra-vesical pressure measured in a standardized way
Round Belly Sign | At the time of CT examination
  Increased ratio of anteroposterior/transverse diameter of the abdomen (ratio >0.80), measured at the level where left renal vein crosses the aorta, excluding subcutaneous fat.

SECONDARY OUTCOMES:
Narrowing of abdomen large veins | At the time of CT examination
  Defined as a slit-like appearance of less than 3 mm
Elevation of the diaphragm | At the time of CT examination
  Defined as dome of diaphragm reaching the 10th thoracic vertebral body or above
Compression or displacement of solid abdominal viscera | At the time of CT examination
  Presence of contour deformity
Bowel wall thickening with contrast enhancement | At the time of CT examination
  Defined as a thickness of 3 mm or greater with contrast enhancement
Bilateral inguinal herniation | At the time of CT examination
  Bilateral inguinal herniation, if not present on a previous imaging examination
Increase of the peritoneal/abdominal ratio | At the time of CT examination
  Increase of the peritoneal/abdominal height ratio (ratio > 0,5). Peritoneal compartment height is measured from posterior third duodenum wall on the median line to the abdominal anterior wall. Abdominal compartment height is measured at the same level, excluding subcutaneous fat.
Semi lunar line distension | At the time of CT examination
  The longer length between transverse abdominis muscle and rectus abdominis muscle in millimeter
Concavity of the upper side of the para renal fascia | At the time of CT examination
  Concave deformity of the upper side of the para renal fascia, with or without renal deformity or displacement
Abdominal Compartment Syndrome (ACS) | From the time of inclusion to 28 days after
  Incidence of ACS in included patients, defined by a sustained intra abdominal hypertension above 20 mmHg and a multiple organ failure due to the raise of the intra abdominal pressure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luckianow GM, Ellis M, Governale D, Kaplan LJ. Abdominal compartment syndrome: risk factors, diagnosis, and current therapy. Crit Care Res Pract. 2012;2012:908169. doi: 10.1155/2012/908169. Epub 2012 Jun 7. PMID 22720147
- [Background] Malbrain ML, De Keulenaer BL, Oda J, De Laet I, De Waele JJ, Roberts DJ, Kirkpatrick AW, Kimball E, Ivatury R. Intra-abdominal hypertension and abdominal compartment syndrome in burns, obesity, pregnancy, and general medicine. Anaesthesiol Intensive Ther. 2015;47(3):228-40. doi: 10.5603/AIT.a2015.0021. Epub 2015 May 14. PMID 25973659
- [Background] Patel A, Lall CG, Jennings SG, Sandrasegaran K. Abdominal compartment syndrome. AJR Am J Roentgenol. 2007 Nov;189(5):1037-43. doi: 10.2214/AJR.07.2092. PMID 17954637
- [Background] Epelman M, Soudack M, Engel A, Halberthal M, Beck R. Abdominal compartment syndrome in children: CT findings. Pediatr Radiol. 2002 May;32(5):319-22. doi: 10.1007/s00247-001-0569-3. Epub 2002 Feb 15. PMID 11956717
- [Background] Al-Bahrani AZ, Abid GH, Sahgal E, O'shea S, Lee S, Ammori BJ. A prospective evaluation of CT features predictive of intra-abdominal hypertension and abdominal compartment syndrome in critically ill surgical patients. Clin Radiol. 2007 Jul;62(7):676-82. doi: 10.1016/j.crad.2006.11.006. Epub 2007 May 2. PMID 17556037
- [Background] Malbrain ML, Chiumello D, Cesana BM, Reintam Blaser A, Starkopf J, Sugrue M, Pelosi P, Severgnini P, Hernandez G, Brienza N, Kirkpatrick AW, Schachtrupp A, Kempchen J, Estenssoro E, Vidal MG, De Laet I, De Keulenaer BL; WAKE-Up! Investigators. A systematic review and individual patient data meta-analysis on intra-abdominal hypertension in critically ill patients: the wake-up project. World initiative on Abdominal Hypertension Epidemiology, a Unifying Project (WAKE-Up!). Minerva Anestesiol. 2014 Mar;80(3):293-306. Epub 2013 Dec 12. PMID 24603146
- [Background] Atema JJ, van Buijtenen JM, Lamme B, Boermeester MA. Clinical studies on intra-abdominal hypertension and abdominal compartment syndrome. J Trauma Acute Care Surg. 2014 Jan;76(1):234-40. doi: 10.1097/TA.0b013e3182a85f59. No abstract available. PMID 24368386
- [Background] Wu J, Zhu Q, Zhu W, Chen W, Wang S. [Computed tomographic features of abdominal compartment syndrome complicated by severe acute pancreatitis]. Zhonghua Yi Xue Za Zhi. 2014 Nov 25;94(43):3378-81. Chinese. PMID 25622665
- [Background] Iyer D, Rastogi P, Aneman A, D'Amours S. Early screening to identify patients at risk of developing intra-abdominal hypertension and abdominal compartment syndrome. Acta Anaesthesiol Scand. 2014 Nov;58(10):1267-75. doi: 10.1111/aas.12409. PMID 25307712
- [Background] De Waele JJ, Ejike JC, Leppaniemi A, De Keulenaer BL, De Laet I, Kirkpatrick AW, Roberts DJ, Kimball E, Ivatury R, Malbrain ML. Intra-abdominal hypertension and abdominal compartment syndrome in pancreatitis, paediatrics, and trauma. Anaesthesiol Intensive Ther. 2015;47(3):219-27. doi: 10.5603/AIT.a2015.0027. Epub 2015 May 14. PMID 25973660
- [Background] Wachsberg RH, Sebastiano LL, Levine CD. Narrowing of the upper abdominal inferior vena cava in patients with elevated intraabdominal pressure. Abdom Imaging. 1998 Jan-Feb;23(1):99-102. doi: 10.1007/s002619900295. PMID 9437074
- [Background] Hong JJ, Cohn SM, Perez JM, Dolich MO, Brown M, McKenney MG. Prospective study of the incidence and outcome of intra-abdominal hypertension and the abdominal compartment syndrome. Br J Surg. 2002 May;89(5):591-6. doi: 10.1046/j.1365-2168.2002.02072.x. PMID 11972549
- [Background] Malbrain ML, Cheatham ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Johansson K, Kolkman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. I. Definitions. Intensive Care Med. 2006 Nov;32(11):1722-32. doi: 10.1007/s00134-006-0349-5. Epub 2006 Sep 12. PMID 16967294
- [Background] Holodinsky JK, Roberts DJ, Ball CG, Blaser AR, Starkopf J, Zygun DA, Stelfox HT, Malbrain ML, Jaeschke RC, Kirkpatrick AW. Risk factors for intra-abdominal hypertension and abdominal compartment syndrome among adult intensive care unit patients: a systematic review and meta-analysis. Crit Care. 2013 Oct 21;17(5):R249. doi: 10.1186/cc13075. PMID 24144138